CLINICAL TRIAL: NCT05236270
Title: CATCH-UP Vaccines: Extension of Community - Engaged Approaches to Testing in Community and Healthcare Settings for Underserved Populations
Brief Title: CATCH-UP Vaccines: Engaged Approaches to Testing in Community/Healthcare Settings for the Underserved (COVID-19)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 13436; 3U54GM104938-09S3 (NIH)
Record Dates: First submitted 2022-02-01; First posted 2022-02-11 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: COVID-19; Vaccine Refusal
Keywords: COVID-19 Vaccine Hesitancy; MOST (multiphase optimization strategy)
MeSH Terms: conditions — COVID-19; Vaccination Refusal | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Interventions will address three primary areas to improve vaccination uptake: (1) process (text messages); (2) teachable moment messaging (motivational interviewing); and (3) barrier elicitation and reduction (electronic survey with tailored questions/prompts). In a factorial research design, two or more independent variables are concurrently examined within the same trial. The three factors are crossed with one another to create a total of eight experimental conditions. An equal number of sites are randomly assigned to each condition, using a random number generator.
Masking Description: Investigators who are providing the intervention and conducting analysis will be masked to study assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Condition 1 (No Intervention): Participants will not receive a text message notifying participants about COVID-19 vaccine availability, standard interpretation of serology SARS-CoV-2 antibody results with COVID-19 vaccination discussion, and an attention control educational message.
- Condition 2 (Experimental): Participants will not receive a text message notifying participants about COVID-19 vaccine availability, standard interpretation of serology SARS-CoV-2 antibody results with COVID-19 vaccination discussion, and an educational message about COVID-19 vaccines.
  Interventions: Behavioral: Electronic Educational Message with Tailored Questions/Prompts
- Condition 3 (Experimental): Patients will not receive a text message notifying participants about COVID-19 vaccine availability, motivational interviewing about serology SARS-CoV-2 antibody results with COVID-19 vaccination discussion, and an attention control educational message.
  Interventions: Behavioral: Motivational Interviewing
- Condition 4 (Experimental): Patients will not receive a text message notifying participants about COVID-19 vaccine availability, motivational interviewing about serology SARS-CoV-2 antibody results with vaccination discussion, and an educational message about COVID-19 vaccines.
  Interventions: Behavioral: Motivational Interviewing; Behavioral: Electronic Educational Message with Tailored Questions/Prompts
- Condition 5 (Experimental): Patients will receive a text message notifying participants about COVID-19 vaccine availability, motivational interviewing about serology SARS-CoV-2 antibody results with vaccination discussion, and an educational message about COVID-19 vaccines.
  Interventions: Behavioral: Text Message; Behavioral: Motivational Interviewing; Behavioral: Electronic Educational Message with Tailored Questions/Prompts
- Condition 6 (Experimental): Patients will receive a text message notifying participants about COVID-19 vaccine availability, motivational interviewing about serology SARS-CoV-2 antibody results with vaccination discussion, and an attention control educational message.
  Interventions: Behavioral: Text Message; Behavioral: Motivational Interviewing
- Condition 7 (Experimental): Patients will receive a text message notifying participants about COVID-19 vaccine availability, standard interpretation of serology SARS-CoV-2 antibody results with COVID-19 vaccination discussion, and an attention control educational message.
  Interventions: Behavioral: Text Message
- Condition 8 (Experimental): Patients will receive a text message notifying participants about COVID-19 vaccine availability, standard interpretation of serology SARS-CoV-2 antibody results with COVID-19 vaccination discussion, and an educational message about COVID-19 vaccines.
  Interventions: Behavioral: Text Message; Behavioral: Electronic Educational Message with Tailored Questions/Prompts

INTERVENTIONS:
Behavioral: Text Message — Participants will be randomized to receive or not receive a text message encouraging COVID-19 vaccine uptake.
  Arms: Condition 5; Condition 6; Condition 7; Condition 8
Behavioral: Motivational Interviewing — Participants will be randomized to receive either motivational interviewing when receiving SARS-CoV-2 antibody test results or standard interpretation of antibody results.
  Arms: Condition 3; Condition 4; Condition 5; Condition 6
Behavioral: Electronic Educational Message with Tailored Questions/Prompts — Participants will be randomized to receive either an electronic educational message tailored to their COVID-19 vaccine concerns and vaccine status or an attention control message about overall healthy choices.
  Arms: Condition 2; Condition 4; Condition 5; Condition 8

SUMMARY:
Oklahoma has high COVID-19 incidence, particularly among underserved minority and rural Oklahomans. Oklahoman's are also reporting SARS-CoV-2 vaccine hesitancy and signs of slowing vaccine uptake, with increased hesitancy among American Indian and rural populations. The project aims to work with ongoing community testing events to implement interventions to improve vaccine uptake among Oklahoma's underserved populations.

DETAILED DESCRIPTION:
This proposal unites academic and community partners to solve a dire need for SARS-CoV-2 vaccine uptake in rural, underserved minority, and at-risk populations. Oklahoma has high COVID-19 incidence, high vaccine hesitancy, and signs of a slowing SARS-CoV-2 vaccine uptake. Oklahoma's cumulative incidence is higher in rural compared to urban counties. AI people have a higher incidence of COVID-19 compared to white populations in Oklahoma. Despite high incidence, as of April 2021, an estimated 54% of Oklahomans who have not yet been vaccinated reported unwillingness to receive the SARS-CoV-2 vaccine. Vaccine hesitancy was even greater in AI people (62%). The most commonly reported concerns are vaccine side effects and safety (30%). Despite early progress in disseminating vaccines in Oklahoma, all signs point to waning interest in receiving a vaccine, with many vaccine clinics unable to fill all available slots, particularly in tribal clinics and rural areas. This proposal is an extension of the Oklahoma Shared Clinical Translational Resources (OSCTR) project CATCH-UP (Community-engaged Approaches to Testing in Community and Healthcare settings for Underserved Populations) in partnership with community organizations who work with underserved minority and rural populations. This project will build on existing strengths and infrastructure to improve SARS-CoV-2 vaccine uptake in these highly susceptible populations. The goal of the project is to pilot interventions to improve awareness and uptake of COVID-19 vaccination. The project aims to work with CATCH-UP community events to implement interventions to improve vaccine uptake among Oklahoma's underserved populations. To do so, the proposed study employs a multiphase optimization strategy (MOST). The proposed study uses the preparation and optimization phases of the MOST framework across the following aims: 1) Identify SARS-CoV-2 vaccination barriers/facilitators and assess acceptability and feasibility of a suite of evidence-based vaccine intervention strategies among Oklahoma's rural, minority, and high-risk populations to inform a targeted multicomponent intervention; and 2) Develop and optimize a multicomponent intervention to improve SARS-CoV-2 vaccination among Oklahoman's seeking SARS-CoV-2 testing at CATCH-UP testing events. Investigators will conduct a pilot of these interventions based on community input, which will be evaluated for inclusion in a future, full-scale implementation study.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older
2. Must be eligible to receive a COVID-19 vaccine dose at the time of consent based on the following criteria:

   a. Eligible for one bivalent mRNA vaccine i. No previous doses of any COVID-19 vaccine ii. At least 8 weeks since a previous vaccine dose of any manufacturer b. Eligible for second bivalent mRNA vaccine i. Adults 65 year of age and older can receive one additional bivalent mRNA vaccine at least 4 months after the first dose of a bivalent mRNA vaccine.

   ii. Those who are immunocompromised can receive one additional bivalent mRNA vaccine at least 2 months after the first dose of a bivalent mRNA vaccine.
3. Ability to read and speak English

Exclusion Criteria:

1. Those who have received all eligible doses of any approved COVID-19 vaccine.
2. Those with active COVID-19 disease (either through self-reported positive test within the last 10 days or viral test at the event if available).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith A James, MD, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- Oklahoma Clinical and Translational Science Institute, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Escoffery C, Riehman K, Watson L, Priess AS, Borne MF, Halpin SN, Rhiness C, Wiggins E, Kegler MC. Facilitators and Barriers to the Implementation of the HPV VACs (Vaccinate Adolescents Against Cancers) Program: A Consolidated Framework for Implementation Research Analysis. Prev Chronic Dis. 2019 Jul 3;16:E85. doi: 10.5888/pcd16.180406. PMID 31274411
- [Background] Garbutt JM, Dodd S, Walling E, Lee AA, Kulka K, Lobb R. Barriers and facilitators to HPV vaccination in primary care practices: a mixed methods study using the Consolidated Framework for Implementation Research. BMC Fam Pract. 2018 May 7;19(1):53. doi: 10.1186/s12875-018-0750-5. PMID 29734944
- [Background] Jacobs-Wingo JL, Espey DK, Groom AV, Phillips LE, Haverkamp DS, Stanley SL. Causes and Disparities in Death Rates Among Urban American Indian and Alaska Native Populations, 1999-2009. Am J Public Health. 2016 May;106(5):906-14. doi: 10.2105/AJPH.2015.303033. Epub 2016 Feb 18. PMID 26890168
- [Background] Nguyen KH, Srivastav A, Razzaghi H, Williams W, Lindley MC, Jorgensen C, Abad N, Singleton JA. COVID-19 Vaccination Intent, Perceptions, and Reasons for Not Vaccinating Among Groups Prioritized for Early Vaccination - United States, September and December 2020. MMWR Morb Mortal Wkly Rep. 2021 Feb 12;70(6):217-222. doi: 10.15585/mmwr.mm7006e3. PMID 33571174
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Proctor EK, Landsverk J, Aarons G, Chambers D, Glisson C, Mittman B. Implementation research in mental health services: an emerging science with conceptual, methodological, and training challenges. Adm Policy Ment Health. 2009 Jan;36(1):24-34. doi: 10.1007/s10488-008-0197-4. Epub 2008 Dec 23. PMID 19104929
- [Background] Raifman MA, Raifman JR. Disparities in the Population at Risk of Severe Illness From COVID-19 by Race/Ethnicity and Income. Am J Prev Med. 2020 Jul;59(1):137-139. doi: 10.1016/j.amepre.2020.04.003. Epub 2020 Apr 27. No abstract available. PMID 32430225
- [Derived] Janitz AE, Neil JM, Bray LA, Jervis LL, Ross L, Campbell JE, Doescher MP, Spicer PG, Williams ML, Lopez AK, Uribe-Frias CA, Chen S, James JA, VanWagoner TM. CATCH-UP vaccines: protocol for a randomized controlled trial using the multiphase optimization strategy (MOST) framework to evaluate education interventions to increase COVID-19 vaccine uptake in Oklahoma. BMC Public Health. 2023 Jun 14;23(1):1146. doi: 10.1186/s12889-023-16077-w. PMID 37316843
- See also: COVID Data Tracker — https://covid.cdc.gov/covid-data-tracker/
- See also: COVID-19 Vaccination Communication: Applying Behavioral and Social Science to Address Vaccine Hesitancy and Foster Vaccine Confidence — https://obssr.od.nih.gov/wp-content/uploads/2020/12/COVIDReport_Final.pdf
- See also: Low-Income and Communities of Color at Higher Risk of Serious Illness if Infected with Coronavirus — https://www.kff.org/disparities-policy/issue-brief/low-income-and-communities-of-color-at-higher-risk-of-serious-illness-if-infected-with-coronavirus/
- See also: CPSTF Findings for Increasing Vaccination — https://www.thecommunityguide.org/content/task-force-findings-increasing-vaccination

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from March 25, 2022 through June 27, 2023 from 21 sites across Oklahoma. Recruitment sites included community events, employee wellness events at healthcare facilities, and conferences.
Pre-assignment Details: After participants provided informed consent and HIPAA authorization, participants were randomized to a treatment condition.
Period: Overall Study
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8
Started | 42 | 42 | 35 | 35 | 42 | 31 | 41 | 44
Completed | 39 | 40 | 35 | 35 | 40 | 31 | 40 | 41
Not Completed | 3 | 2 | 0 | 0 | 2 | 0 | 1 | 3
Not completed — Lost to Follow-up | 3 | 2 | 0 | 0 | 2 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8 | Total
Number analyzed (Participants) | 42 | 42 | 35 | 35 | 42 | 31 | 41 | 44 | 312
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (12.5) | 47.0 (14.5) | 52.4 (13.4) | 46.8 (14.3) | 44.7 (14.2) | 47.1 (12.8) | 44.4 (14.4) | 43.3 (14.4) | 46.0 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Information on sex was missing for 8 participants across treatment groups.
  Participants
    number analyzed (Participants) | 40 | 41 | 35 | 33 | 41 | 30 | 41 | 43 | 304
    Female | 27 | 32 | 31 | 27 | 32 | 25 | 31 | 34 | 239
    Male | 13 | 9 | 4 | 6 | 9 | 5 | 10 | 9 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 3 | 1 | 5 | 3 | 6 | 5 | 31
  Not Hispanic or Latino | 36 | 37 | 32 | 32 | 36 | 27 | 34 | 37 | 271
  Unknown or Not Reported | 2 | 1 | 0 | 2 | 1 | 1 | 1 | 2 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 0 | 2 | 1 | 3 | 3 | 3 | 17
  Asian | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 1 | 0 | 5 | 5 | 5 | 2 | 24
  White | 32 | 32 | 32 | 31 | 28 | 20 | 28 | 34 | 237
  More than one race | 1 | 2 | 1 | 0 | 2 | 2 | 3 | 1 | 12
  Unknown or Not Reported | 4 | 1 | 1 | 2 | 5 | 1 | 2 | 3 | 19
Region of Enrollment [Number; unit: participants]
  United States | 42 | 42 | 35 | 35 | 42 | 31 | 41 | 44 | 312

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Plan to Receive a COVID-19 Vaccine Post-intervention
Description: Investigators will measure this with the question "How likely are you to get an approved COVID-19 vaccine?" and "If you have received 1 dose of the Janssen vaccine or 2 doses of the Moderna or Pfizer vaccine, how likely are you to get an approved booster shot?" We will compare intention to receive a COVID-19 vaccine or booster among those receiving the interventions compared to those not receiving the intervention
Time Frame: Baseline to Post-Intervention Survey (approximately 15-30 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8
Number analyzed (Participants) | 42 | 42 | 35 | 35 | 42 | 31 | 41 | 44
Participants | 19 | 24 | 19 | 21 | 24 | 19 | 23 | 16

2. Secondary Outcome: Percentage of Participants Who Self-report COVID-19 Vaccine Uptake
Description: The secondary outcome will be vaccine uptake, including self-report of receiving an initial dose of any approved vaccine, two doses of Pfizer or Moderna vaccines, or a booster of any approved vaccine.
Time Frame: Baseline to Month 2
Population: Analysis includes participants who completed the 60-day follow-up survey (n=47)
Measure: Count of Participants; unit: Participants
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8
Number analyzed (Participants) | 7 | 5 | 4 | 5 | 9 | 3 | 10 | 4
Participants | 2 | 1 | 0 | 0 | 2 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the primary study visit, which lasted approximately 30 minutes.
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42 | 0/35 | 0/35 | 0/42 | 0/31 | 0/41 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/35 | 0/35 | 0/42 | 0/31 | 0/41 | 0/44
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/35 | 0/35 | 0/42 | 0/31 | 0/41 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT05236270/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT05236270/ICF_001.pdf